CLINICAL TRIAL: NCT04957758
Title: A Phase 2, Multicenter, Randomized, Controlled, Double-Masked, Clinical Trial to Evaluate the Efficacy and Safety of OC-01 (Varenicline) Nasal Spray in Subjects With Neurotrophic Keratopathy (the Olympia Study)
Brief Title: Phase 2 Clinical Trial to Evaluate OC-01 Nasal Spray in Subjects With Neurotrophic Keratopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPP-102
Record Dates: First submitted 2021-06-28; First posted 2021-07-12 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-03

CONDITIONS: Neurotrophic Keratopathy
MeSH Terms: interventions — Varenicline; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OC-01 (varenicline) nasal spray, 1.2 mg/mL (Active Comparator): OC-01 (varenicline) nasal spray, 1.2 mg/mL
  Interventions: Drug: OC-01 (varenicline) nasal spray 1.2 mg/ml
- Placebo (vehicle control) nasal spray (Placebo Comparator): Placebo (vehicle control) nasal spray
  Interventions: Drug: Placebo (vehicle) nasal spray

INTERVENTIONS:
Drug: OC-01 (varenicline) nasal spray 1.2 mg/ml — OC-01
  Arms: OC-01 (varenicline) nasal spray, 1.2 mg/mL
Drug: Placebo (vehicle) nasal spray — Placebo (vehicle)
  Arms: Placebo (vehicle control) nasal spray

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of OC-01 (varenicline) nasal spray as compared to placebo nasal spray for mean change from baseline in corneal fluorescein staining in subjects with Stage 1 (corneal epithelial hyperplasia/punctate keratopathy) neurotrophic keratopathy (NK) in one or both eyes.

DETAILED DESCRIPTION:
Protocol OPP-102 is a Phase 2, multicenter, randomized, controlled, double- masked study designed to evaluate the safety and efficacy of OC-01 (varenicline) nasal spray in subjects with NK. Approximately 100 subjects at least 18 years of age with a physicians' diagnosis of Stage 1 NK as defined by the Mackie Criteria and meeting all other study eligibility criteria will be randomized 1:1 and will receive OC-01 (varenicline)/ nasal spray or placebo nasal spray for 8 weeks three times daily (TID) as follows:

* OC-01 (varenicline) nasal spray, 1.2 mg/mL
* Placebo (vehicle control) nasal spray All doses will be delivered as a 50 microliter (µL) nasal spray.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age at Visit 1.
2. Patients with Stage 1 (corneal epithelial hyperplasia/punctate keratopathy) NK in one or both eyes, as defined by the Mackie Criteria.
3. Evidence of decreased corneal sensitivity (≤ 4 cm using the Cochet-Bonnet aesthesiometer) in at least 1 corneal quadrant.
4. Schirmer's test without anesthesia ≥3 mm/ 5 minutes in the affected eye.
5. If a female is of childbearing potential, they must: use an acceptable means of birth control (acceptable methods of contraception include hormonal - oral, implantable, injectable, or transdermal contraceptives, mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom, IUD, or surgical sterilization of partner), and have a negative urine pregnancy test on Day 1.

Exclusion Criteria:

1. Have Stage 2 or Stage 3 NK affecting one or both eyes.
2. Have ocular graft versus host disease or Stevens-Johnson syndrome.
3. Have any active ocular infection (COVID-19 conjunctivitis, bacterial, viral, fungal, or protozoal) or active ocular inflammation not related to NK in the affected eye.
4. Be currently receiving autologous serum tears, amniotic membrane, cenegermin, fresh frozen plasma or cord blood derivative tears.
5. Have severe blepharitis and/or severe meibomian gland disease in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Dothan Alabama, Dothan, Alabama
  - Irvine, California, Irvine, California
  - Los Angeles California, Los Angeles, California
  - Mission Hills California, Mission Hills, California
  - Aurora Colorado, Aurora, Colorado
  - Littleton, Colorado, Littleton, Colorado
  - Longmont, Colorado, Longmont, Colorado
  - Danbury, Connecticut, Danbury, Connecticut
  - Brandon Florida, Brandon, Florida
  - Brandon, Florida, Brandon, Florida
  - Jacksonville Florida, Jacksonville, Florida
  - Miami Florida, Miami, Florida
  - Atlanta, Georgia, Atlanta, Georgia
  - Hoffman Estates, Illinois, Hoffman Estates, Illinois
  - Urbana Illinois, Urbana, Illinois
  - Union Kentucky, Edgewood, Kentucky
  - Louisville KY, Louisville, Kentucky
  - Bowie, Maryland, Bowie, Maryland
  - Boston Massachusetts, Boston, Massachusetts
  - Kansas City Missouri, Kansas City, Missouri
  - Henderson Nevada, Henderson, Nevada
  - Bloomfield, New Jersey, Bloomfield, New Jersey
  - Dover New Jersey, Dover, New Jersey
  - Babylon New York, Babylon, New York
  - New York NY, New York, New York
  - York, Pennsylvania, York, Pennsylvania
  - Houston Texas, Houston, Texas
  - Katy, Texas, Katy, Texas
  - San Antonio Texas, San Antonio, Texas
  - Lynchburg Virginia, Lynchburg, Virginia
  - Seattle Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OC-01 (Varenicline) Nasal Spray, 1.2 mg/mL | Placebo (Vehicle Control) Nasal Spray
Started | 53 | 60
Completed | 48 | 55
Not Completed | 5 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OC-01 (Varenicline) Nasal Spray, 1.2 mg/mL | Placebo (Vehicle Control) Nasal Spray | Total
Number analyzed (Participants) | 53 | 60 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (14.48) | 61.5 (16.33) | 63.3 (15.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 47 | 88
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 14 | 23
  Not Hispanic or Latino | 44 | 45 | 89
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 47 | 50 | 97
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Corneal Fluorescein staining Score [Mean (Standard Deviation); unit: units on a scale] — Corneal Fluorescein Staining was measured utilizing the Modified Oxford Grading scale. Scores range from a minimum of 0 (no staining) to a maximum of 5. A higher score indicates a worse outcome.
  units on a scale | 2.29 (1.017) | 2.17 (1.028) | 2.23 (1.020)
Best Correct Visual Acuity (Letters) [Mean (Standard Deviation); unit: Number of letters] — Best Corrected Visual Acuity was assessed based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. ETDRS letters score range from 0 to 100 letters at each assessment.
  A higher score in ETDRS letters indicates a better outcome. A positive change from Baseline in ETDRS letter score indicates an improvement in visual acuity.
  Number of letters | 75.4 (14.42) | 75.9 (18.54) | 75.7 (16.61)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Corneal Fluorescein Staining
Description: Corneal Fluorescein Staining was measured utilizing the Modified Oxford Grading scale. Scores range from a minimum of 0 (no staining) to a maximum of 5. A higher score indicates a worse outcome. The study eye is defined as the eye with the worst staining grade (if both eyes are eligible).
Time Frame: 8 weeks
Population: Per Protocol Population included all subjects in the intent to treat (ITT) population that had a baseline corneal fluorescein staining score >=2.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OC-01 (Varenicline) Nasal Spray, 1.2 mg/mL | Placebo (Vehicle Control) Nasal Spray
Number analyzed (Participants) | 37 | 45
score on a scale | -0.6 (0.17) | -0.9 (0.15)

2. Secondary Outcome: Mean Change From Baseline in Visual Acuity at Week 8
Description: Best Corrected Visual Acuity was assessed based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. ETDRS letters score range from 0 to 100 letters at each assessment.
  A higher score in ETDRS letters indicates a better outcome. A positive change from Baseline in ETDRS letter score indicates an improvement in visual acuity.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OC-01 (Varenicline) Nasal Spray, 1.2 mg/mL | Placebo (Vehicle Control) Nasal Spray
Number analyzed (Participants) | 37 | 45
score on a scale | 0.6 (1.15) | 1.5 (1.03)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected at the time of informed consent until the last study visit at 6 months.
Description: Participant population in the Adverse Events section is the safety population. There was 1 subject that was randomized to the placebo group, however was enrolled in error and not treated. Therefore total number of subjects enrolled is 113 but total treated is 112. Additionally, subjects were analyzed based on randomization, however 1 subject in the placebo group received an active treatment kit so therefore total number randomized to OC-01 is 53 but total treated is 54.
Arm/Group | OC-01 (Varenicline) Nasal Spray, 1.2 mg/mL | Placebo (Vehicle Control) Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/58
Serious Adverse Events (participants affected / at risk) | 5/54 | 3/58
Other Adverse Events (participants affected / at risk) | 39/54 | 34/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OC-01 (Varenicline) Nasal Spray, 1.2 mg/mL (N=54) | Placebo (Vehicle Control) Nasal Spray (N=58)
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Infective Exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OC-01 (Varenicline) Nasal Spray, 1.2 mg/mL (N=54) | Placebo (Vehicle Control) Nasal Spray (N=58)
Corneal Dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Asthenopia (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Corneal Degeneration (Eye disorders) | 1 | 0
Conjunctivochalasis (Eye disorders) | 0 | 1
Corneal epithelium defect (Eye disorders) | 4 | 1
Corneal erosion (Eye disorders) | 1 | 0
Corneal neovascularisation (Eye disorders) | 0 | 1
Corneal Opacity (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Dry Eye (Eye disorders) | 1 | 2
Erythema of eyelid (Eye disorders) | 0 | 1
Eye Discharge (Eye disorders) | 0 | 1
Eye Irritation (Eye disorders) | 2 | 1
Eye Pain (Eye disorders) | 2 | 1
Lacrimation Increased (Eye disorders) | 1 | 0
Meibomian Gland Dysfunction (Eye disorders) | 1 | 1
Ocular Hyperaemia (Eye disorders) | 0 | 2
Punctate Keratitis (Eye disorders) | 0 | 2
Vision Blurred (Eye disorders) | 0 | 1
Visual Acuity Reduced (Eye disorders) | 0 | 1
Vitreous Floaters (Eye disorders) | 0 | 1
Disease Progression (General disorders) | 0 | 1
Pain (General disorders) | 0 | 3
Conjunctivitis (General disorders) | 0 | 1
Erythema of eyelid (Eye disorders) | 1 | 0
Eye Swelling (General disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Instillation Site Exfoliation (General disorders) | 0 | 1
Instillation Site Irritation (General disorders) | 4 | 2
Hypersensitivity (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis escherichia coli (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Herpes Zoster (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Heart Rate Increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1
Cervical Radiculopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Migraine (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Hypertonic Bladder (Renal and urinary disorders) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Nasal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 30 | 6
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Trichorrhexis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT04957758/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT04957758/SAP_002.pdf